CLINICAL TRIAL: NCT05190029
Title: Early Craniosacral and Primitive Reflex Assessment in Infant Neurodevelopment.
Brief Title: Craniosacral Test and Primitive Reflexes in Infant Neurodevelopment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica Gema Leon (Other)
Responsible Party: Principal Investigator, GEMA LEÓN BRAVO, Principal Investigator, Clinica Gema Leon
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ART-GLB-PRIMITIVE REFLEXES
Record Dates: First submitted 2021-12-15; First posted 2022-01-13 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: Child Development Disorder
Keywords: primitive reflexes; craniosacral disfunctions; neurodevelopment; childhood; early diagnosis; screening
MeSH Terms: conditions — Developmental Disabilities; Disease

STUDY DESIGN:
Intervention Model Description: 120 children aged 3 to 8 years from a school in Córdoba (Spain). Subjects of both sexes were included and were divided into two groups according to age ranges: 3 to 6 years and 6 to 8 years.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Complete sample (Experimental): Group of 120 children evaluated by craniosacral therapy for cranial blocks and primitive reflexes.
  Interventions: Diagnostic Test: Series of questions to parents of children in a virtual form.; Other: Intervention by teachers; Procedure: Physiotherapeutic evaluation

INTERVENTIONS:
Diagnostic Test: Series of questions to parents of children in a virtual form. — A questionnaire of 5 questions was provided in an online format addressed to the parents or legal representatives of each child. These questions were related to the child's own aspects (behavioral, psychomotor and cognitive parameters), as well as parameters oriented to the mother (pregnancy and childbirth).
Other: Intervention by teachers — The school teachers examined neurobehavioral aspects of the students using the "Battelle Developmental Inventory" (BDI), which assesses five areas of development (personal/social, adaptive, motor, communicative and cognitive) between 2 and 8 years of age. The results are assigned in age-adjusted percentages, classified as: low (0-50%), normal (50-80%) and high (80-100%). Low and high values are considered impairments in one or more of the evaluated areas.
Procedure: Physiotherapeutic evaluation — A physiotherapeutic evaluation of the state of the RP and craniosacral system was performed according to the method of Andrzej Pilat and John E. Upledger.
  The 14 primitive reflexes explored were: Moro reflex, cervical asymmetric, supine labyrinthine tonic, prone labyrinthine tonic, palmar grasp, plantar grasp, lateral trunk propulsion, parachute, Galant, search, cervical symmetric, Babinski, cochleo-palpebral and acoustic. These reflexes were considered as: inactive (0), or active (1).
  In the evaluation of the craniosacral system, the following parameters were explored: dura mater sway, frontal bone, parietal bones, temporal bones, temporomandibular joint and sphenoid bone. These parameters were considered as: normal (0), or blockage (1).

SUMMARY:
Question(s): Can active primitive reflexes (APR) and cranial blocks (CB) in healthy children interfere with neurological balance causing psycho-behavioral and cognitive dysfunctions? Design: Cross-sectional and descriptive study analyzing perinatal, neurobehavioral and physiotherapeutic parameters. Participants: School population of both genders (n=120) divided in two groups: 3-6 years old (n=60) and 6-8 years old (n=60). Intervention: Systematic evaluation of the children based on a parent survey, assessment by teachers and physiotherapeutic exploration. Outcome measures: Perinatal (surveyed parents) and neurobehavioral problems (assessed by teachers) were related to the presence of RPA and BC (analyzed by physiotherapeutic exploration).

Key words: primitive reflexes, craniosacral disfunctions, neurodevelopment, childhood, early diagnosis, screening.

DETAILED DESCRIPTION:
Primitive reflexes (PR) are indispensable for the survival of the individual in the early stages of life. PR are necessary for a coordinated response to sensory stimuli during the period of cortical immaturity until the maturation of the central nervous system (CNS). However, PR must be gradually abolished as the subject's development proceeds, allowing for voluntary and functional movement responses. This process of PR abolition is due to the synaptic plasticity of the CNS. Persistent ROP can be identified by means of a systematic neurological examination. On the other hand, through craniosacral exploration, blockages in the craniosacral system can be evidenced; under physiological conditions, this system seeks to balance the mobility of membranes and cranial sutures, based on the coordinated movement of the cranial bones and the sacrum. If neurological homeostasis is disturbed in the child after diagnosing possible BC, this could manifest in the persistence of RPA and/or vice versa.

Observation of the child's different behavioral patterns in social and emotional areas, as well as his or her physical and psychological capacities, could help to detect early possible alterations in the onset of neurodevelopment. Such detection is essential for the health professional to be able to establish an appropriate treatment.

The aim of this study is to detect early infant neurodevelopmental dysfunctions and their possible relationship with RPA and/or BC in apparently healthy children.

Therefore, the research questions of this study were:

1. Are RPA and/or BC related to child neurodevelopmental disturbances?
2. In relation to the previous question, by means of the systematic evaluation of RPA and BC could children with neurodevelopmental disorders be identified in order to treat them early?

Design A cross-sectional, observational and descriptive study was conducted in a school population.

Participants, therapists, centers A total of 120 children between 3 and 8 years of age from a school in Córdoba (Spain) were evaluated. Subjects of both sexes were included and were divided into two groups according to age ranges: 3 to 6 years and 6 to 8 years. The neurodevelopmental assessment was made taking into account the growth stages standardized by the WHO.

Prior approval was obtained from the Research Ethics Committee of Córdoba for the present study. The harmonized tripartite standards of the Helsinki declaration, the Biomedical Research Law (Law 14/2007), and the Organic Law on Personal Data Protection (Organic Law 3/2018) were respected at all times. The application of tests and data collection for the research was performed within the facilities of the educational institution, with the collaboration of the teachers and having the due authorization of the academic director and the parents or legal representatives of the students.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy children
* School group
* Within age range

Exclusion Criteria:

* Children with possible pathologies
* Older than the established age

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-02-05 (Actual)

PRIMARY OUTCOMES:
Series of questions to the children's parents | one week
  A questionnaire of 5 questions in an online format was sent to the parents or legal representatives of each child related to behavioral, psychomotor and cognitive aspects, pregnancy and childbirth.
Teachers' test by means of the "Battelle Development Inventory" (BDI). | Three weeks
  The school teachers examined neurobehavioral aspects of the students using the "Battelle Developmental Inventory" (BDI), which assesses five areas of development (personal/social, adaptive, motor, communicative and cognitive) between 2 and 8 years of age. The results are assigned in age-adjusted percentages, classified as: low (0-50%), normal (50-80%) and high (80-100%). Low and high values are considered impairments in one or more of the evaluated areas.

SECONDARY OUTCOMES:
Craniosacral evaluation of possible cranial blocks | Three weeks
  In the evaluation of the craniosacral system, the following parameters were explored: dura mater sway, frontal bone, parietal bones, temporal bones, temporomandibular joint and sphenoid bone. These parameters were considered as: normal (0), or blockage (1).
Craniosacral evaluation of active primitive reflexes. | Three weeks
  14 primitive reflexes explored were: Moro reflex, cervical asymmetric, supine labyrinthine tonic, prone labyrinthine tonic, palmar prehension, plantar prehension, lateral trunk propulsion, parachute, Galant, search, cervical symmetric, Babinski, cochleo-palpebral and acoustic. These reflexes were considered as: inactive (0), or active (1).

CONTACTS AND LOCATIONS:
Overall Officials: Irene Cantarero, Study Chair, Study Chair — Universidad de Córdoba; Javier Caballero Villarraso, Study Direct, Study Director — Universidad de Córdoba
Locations (1):
- Clinica de Fisioterapia Gema León, Córdoba, Andalusia, Spain

IPD SHARING:
Plan to Share IPD: No
The request for data will be studied and considered upon justified request.

REFERENCES:
- [Background] Pecuch A, Gieysztor E, Telenga M, Wolanska E, Kowal M, Paprocka-Borowicz M. Primitive Reflex Activity in Relation to the Sensory Profile in Healthy Preschool Children. Int J Environ Res Public Health. 2020 Nov 6;17(21):8210. doi: 10.3390/ijerph17218210. PMID 33172138
- [Background] Pecuch A, Gieysztor E, Wolanska E, Telenga M, Paprocka-Borowicz M. Primitive Reflex Activity in Relation to Motor Skills in Healthy Preschool Children. Brain Sci. 2021 Jul 23;11(8):967. doi: 10.3390/brainsci11080967. PMID 34439585
- [Background] Gieysztor EZ, Choinska AM, Paprocka-Borowicz M. Persistence of primitive reflexes and associated motor problems in healthy preschool children. Arch Med Sci. 2018 Jan;14(1):167-173. doi: 10.5114/aoms.2016.60503. Epub 2016 Jun 13. PMID 29379547
- [Background] Bob P, Konicarova J, Raboch J. Disinhibition of Primitive Reflexes in Attention Deficit and Hyperactivity Disorder: Insight Into Specific Mechanisms in Girls and Boys. Front Psychiatry. 2021 Nov 8;12:430685. doi: 10.3389/fpsyt.2021.430685. eCollection 2021. PMID 34819879
- [Background] Konicarova J, Bob P, Raboch J. Persisting primitive reflexes in medication-naive girls with attention-deficit and hyperactivity disorder. Neuropsychiatr Dis Treat. 2013;9:1457-61. doi: 10.2147/NDT.S49343. Epub 2013 Sep 20. PMID 24092983
- [Background] Melillo R, Leisman G, Mualem R, Ornai A, Carmeli E. Persistent Childhood Primitive Reflex Reduction Effects on Cognitive, Sensorimotor, and Academic Performance in ADHD. Front Public Health. 2020 Nov 17;8:431835. doi: 10.3389/fpubh.2020.431835. eCollection 2020. PMID 33282806
- [Background] Sohn M, Ahn Y, Lee S. Assessment of Primitive Reflexes in High-risk Newborns. J Clin Med Res. 2011 Dec;3(6):285-90. doi: 10.4021/jocmr706w. Epub 2011 Nov 10. PMID 22393339
- [Background] Marin Gabriel MA, Olza Fernandez I, Malalana Martinez AM, Gonzalez Armengod C, Costarelli V, Millan Santos I, Fernandez-Canadas Morillo A, Perez Riveiro P, Lopez Sanchez F, Garcia Murillo L. Intrapartum synthetic oxytocin reduce the expression of primitive reflexes associated with breastfeeding. Breastfeed Med. 2015 May;10(4):209-13. doi: 10.1089/bfm.2014.0156. Epub 2015 Mar 18. PMID 25785487
- [Background] Vreeling FW, Verhey FR, Houx PJ, Jolles J. Primitive reflexes in Parkinson's disease. J Neurol Neurosurg Psychiatry. 1993 Dec;56(12):1323-6. doi: 10.1136/jnnp.56.12.1323. PMID 8270937
- [Background] Futagi Y, Toribe Y, Suzuki Y. The grasp reflex and moro reflex in infants: hierarchy of primitive reflex responses. Int J Pediatr. 2012;2012:191562. doi: 10.1155/2012/191562. Epub 2012 Jun 11. PMID 22778756
- [Background] Gieysztor E, Pecuch A, Kowal M, Borowicz W, Paprocka-Borowicz M. Pelvic Symmetry Is Influenced by Asymmetrical Tonic Neck Reflex during Young Children's Gait. Int J Environ Res Public Health. 2020 Jul 2;17(13):4759. doi: 10.3390/ijerph17134759. PMID 32630679
- [Background] Huber SJ, Paulson GW. Relationship between primitive reflexes and severity in Parkinson's disease. J Neurol Neurosurg Psychiatry. 1986 Nov;49(11):1298-300. doi: 10.1136/jnnp.49.11.1298. PMID 3794736
- [Background] Niklasson M, Norlander T, Niklasson I, Rasmussen P. Catching-up: Children with developmental coordination disorder compared to healthy children before and after sensorimotor therapy. PLoS One. 2017 Oct 11;12(10):e0186126. doi: 10.1371/journal.pone.0186126. eCollection 2017. PMID 29020061
- [Background] Haller H, Lauche R, Cramer H, Rampp T, Saha FJ, Ostermann T, Dobos G. Craniosacral Therapy for the Treatment of Chronic Neck Pain: A Randomized Sham-controlled Trial. Clin J Pain. 2016 May;32(5):441-9. doi: 10.1097/AJP.0000000000000290. PMID 26340656
- [Background] Wetzler G, Roland M, Fryer-Dietz S, Dettmann-Ahern D. CranioSacral Therapy and Visceral Manipulation: A New Treatment Intervention for Concussion Recovery. Med Acupunct. 2017 Aug 1;29(4):239-248. doi: 10.1089/acu.2017.1222. PMID 28874926
- [Background] Raith W, Marschik PB, Sommer C, Maurer-Fellbaum U, Amhofer C, Avian A, Lowenstein E, Soral S, Muller W, Einspieler C, Urlesberger B. General Movements in preterm infants undergoing craniosacral therapy: a randomised controlled pilot-trial. BMC Complement Altern Med. 2016 Jan 13;16:12. doi: 10.1186/s12906-016-0984-5. PMID 26758035
- [Background] Curtis P, Gaylord SA, Park J, Faurot KR, Coble R, Suchindran C, Coeytaux RR, Wilkinson L, Mann JD. Credibility of low-strength static magnet therapy as an attention control intervention for a randomized controlled study of CranioSacral therapy for migraine headaches. J Altern Complement Med. 2011 Aug;17(8):711-21. doi: 10.1089/acm.2010.0277. Epub 2011 Jul 6. PMID 21732734
- [Background] Mann JD, Faurot KR, Wilkinson L, Curtis P, Coeytaux RR, Suchindran C, Gaylord SA. Craniosacral therapy for migraine: protocol development for an exploratory controlled clinical trial. BMC Complement Altern Med. 2008 Jun 9;8:28. doi: 10.1186/1472-6882-8-28. PMID 18541041
- [Background] Haller H, Lauche R, Sundberg T, Dobos G, Cramer H. Craniosacral therapy for chronic pain: a systematic review and meta-analysis of randomized controlled trials. BMC Musculoskelet Disord. 2019 Dec 31;21(1):1. doi: 10.1186/s12891-019-3017-y. PMID 31892357
- [Background] Ghasemi C, Amiri A, Sarrafzadeh J, Dadgoo M, Jafari H. Comparative study of muscle energy technique, craniosacral therapy, and sensorimotor training effects on postural control in patients with nonspecific chronic low back pain. J Family Med Prim Care. 2020 Feb 28;9(2):978-984. doi: 10.4103/jfmpc.jfmpc_849_19. eCollection 2020 Feb. PMID 32318454
- [Background] Mataran-Penarrocha GA, Castro-Sanchez AM, Garcia GC, Moreno-Lorenzo C, Carreno TP, Zafra MD. Influence of craniosacral therapy on anxiety, depression and quality of life in patients with fibromyalgia. Evid Based Complement Alternat Med. 2011;2011:178769. doi: 10.1093/ecam/nep125. Epub 2011 Jun 15. PMID 19729492